CLINICAL TRIAL: NCT04783662
Title: Study of an Intraoperative Frontal Electroencephalographic Marker of Preoperative Frailty in Patients Over 65 Years of Age for Elective Non-cardiac Surgery.
Brief Title: Intraoperative EEG Marker of Preoperative Frailty in Elderly Patients
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Other Study IDs: 200927001
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2021-01

CONDITIONS: Frailty
Keywords: Frailty; Electroencephalography; Pre operative; Alpha power
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Robust: Patients ≥65 years, undergoing elective non cardiac surgery which Fried phenotype score is equal to 0
  Interventions: Device: Intraoperative frontal electroencephalogram
- Pre Frail: Patients ≥65 years, undergoing elective non cardiac surgery which Fried phenotype score is 1 or 2
  Interventions: Device: Intraoperative frontal electroencephalogram
- Frail: Patients ≥65 years, undergoing elective non cardiac surgery which Fried phenotype score is equal or greater than 3
  Interventions: Device: Intraoperative frontal electroencephalogram

INTERVENTIONS:
Device: Intraoperative frontal electroencephalogram — Intra operative frontal electroencephalogram registration with 1 age adjusted Minimum Anesthetic Concentration of Sevoflurane

SUMMARY:
Frailty is a state of vulnerability, characterized by a loss of mechanisms that maintain homeostasis, determining a lower capacity for recovery in the event of a stressful incident. It is one of the risk factors that increase postoperative adverse outcomes in the elderly population. It has been associated with worse results in different surgical settings, including increased mortality, readmission, referral to specialized care units, increased costs and hospital stay. Currently, there are several instruments for diagnosis and screening of frailty. All of them require time for their execution, an experienced evaluator and an adequate validation in the population in which they are intended to be used. The use of frontal electroencephalography during the intraoperative period has become increasingly popular. It allows the monitoring of brain activity during the administration of anesthetics. Various intraoperative electroencephalographic markers, such as alpha spectral power or total spectrum power, have been associated with factors such as preoperative physical activity, preoperative cognitive level, comorbidities, and postoperative delirium. The objective of this study will be to determine an intraoperative frontal electroencephalographic marker of preoperative frailty in ≥ 65 years patients undergoing general anesthesia with Sevoflurane for non-cardiac surgery.

DETAILED DESCRIPTION:
The world health organization has estimated that the population over 60 years of age will increase exponentially between 2015 and 2050. This change will be more pronounced in developing countries, including Chile. Each year, the number of older people (≥ 65 years) undergoing surgical interventions raises. This is due to a sustained increase in life expectancy, demographic changes, and progress in surgical/anesthetic techniques that allow this population to undergo less invasive procedures. In addition, older patients have a higher risk of postoperative morbidity and mortality compared to younger people.

Frailty is one of the risk factors that increase adverse postoperative outcomes in the elderly population. It is defined as a state of vulnerability or lack of physiological reserve that is characterized by an inadequate resolution of homeostasis after a stressful event. Frailty determines that an event can generate changes in the postoperative state of dependence of these patients; causing a person who was independent prior to surgery to end up requiring assistance with their activities of daily living after it. Frailty has been associated with worse outcomes in different surgical settings, including increased mortality, readmission, referral to specialized care units, increased costs and hospital stay. In addition, preoperative frailty has also been associated with postoperative delirium.

Currently, there are several instruments for the diagnosis and screening of frailty that present good sensitivity and specificity. All of them require time for their execution, an experienced evaluator and adequate validation in the population in which they are intended to be used. Furthermore, with some instruments, specific elements may be required, for example the Handgrip dynamometer for the Fried phenotype. These conditions are not always easy to obtain in the local preoperative setting and the tools are not always adequately validated for non-English speaking populations. Moreover, there is uncertainty regarding which frailty instrument to choose among the dozens described in the literature, and there are time pressures that prevent the addition of more tests or evaluations in the preoperative clinic.

The use of frontal electroencephalography (EEG) during the intraoperative period has become increasingly popular. It is used to obtain a real-time record of brain electrical activity during administration of anesthetics. Interpreting the EEG in the time domain in real time in the operation room is challenging. Therefore, various processed EEG monitors (BIS®, SedLine®) currently clinically used, have incorporated the spectral analysis to their records. The spectrum presents the advantage to show the frequency decomposition of the EEG segment for all frequencies in a given range (usually <30 Hz) by plotting the frequency on the X axis and power on the Y axis. The accumulation of spectra over time is called spectrogram and can be presented graphically on the monitor, where the X-axis represents time, Y axis the decomposition of frequencies, and the Z bar represents the amplitude or power of the different waves. With increasing age there is a decrease in spectral power and alpha wave coherence (8-12 Hz). In addition, decreased alpha spectral power during anesthetic administration has been correlated with preoperative cognitive dysfunction. Recently, preoperative physical activity, the spectral power of the alpha wave and the entire spectral band have been associated with postoperative delirium in the cardio-surgical population. In addition, the spectral power of the alpha wave and broadband power (baseline noise) has been correlated with changes in age and patient comorbidities.

The objective of this study will be to determine an intraoperative frontal electroencephalographic marker of preoperative frailty in a population older than 65 years undergoing general anesthesia with sevoflurane for elective non-cardiac surgery. Our hypothesis is that frail patients (determined by the FRAIL, Clinical Frailty Scale and Fried scales) undergoing general anesthesia with sevofluorane for non-cardiac surgery have a lower alpha spectral power and lower entire spectral band power of the EEG compared to patients of similar age, who are robust, undergoing the same type of surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 65 years of age
* Undergoing elective non-cardiac surgery requiring general anesthesia with Sevoflurane
* American Society of Anesthesiologists Physical Status I to III

Exclusion Criteria:

* Emergency surgery
* Neurosurgical patients
* History of alcohol
* History of recreational psychoactive drug use
* Allergy to anesthetic drugs.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients ≥ 65 years scheduled for elective non-cardiac surgery requiring general anesthesia.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Electroencephalogram Alpha power | 10 minutes after airway intubation
  Frontal electroencephalogram spectral power between 8 - 12 Hz

SECONDARY OUTCOMES:
Electroencephalogram Total power | 10 minutes after airway intubation
  Frontal electroencephalogram spectral power between 0.1 - 35 Hz
Fried Phenotype | During preoperative anesthetic visit
  Frailty assessed with the Fried Phenotype, minimum value: 1 - maximum value: 5, higher scores meaning worse outcomes.
FRAIL scale | During preoperative anesthetic visit
  Frailty assessed with the FRAIL Scale, minimum value: 1 - maximum value: 5, higher scores meaning worse outcomes.
Clinical Frailty Scale (CFS) | During preoperative anesthetic visit
  Frailty assessed with CFS, minimum value: 1(Very fit) - maximum value: 9 (Terminally ill), higher scores meaning worse outcomes.
MiniCog test | During preoperative anesthetic visit
  Screening for cognitive impairment, minimum value: 0 - maximum value: 5, higher scores meaning better outcomes
MOCA (Montreal Cognitive Assessment) test | During preoperative anesthetic visit, if MiniCog is positive for cognitive impairment
  Cognitive evaluation using MOCA (Montreal Cognitive Assessment) test, if MiniCog is positive for cognitive impairment (MiniCog ≤ 2). Minimum value: 0 - maximum value: 30, higher scores meaning better outcomes
Post Anesthesia Care Unit (PACU) Postoperative Delirium | One hour after patient is admitted to PACU
  Confusion Assessment Method for the Intensive Care Unit (CAM-ICU), positive or negative

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Pedemonte, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Hospital Clínico Pontificia Universidad Católica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided
All data will be collected and saved in digital forms. Data may be shared with other researchers with previous authorization from the PI.

REFERENCES:
- [Background] Soreide K, Wijnhoven BP. Surgery for an ageing population. Br J Surg. 2016 Jan;103(2):e7-9. doi: 10.1002/bjs.10071. No abstract available. PMID 26771471
- [Background] Fowler AJ, Abbott TEF, Prowle J, Pearse RM. Age of patients undergoing surgery. Br J Surg. 2019 Jul;106(8):1012-1018. doi: 10.1002/bjs.11148. Epub 2019 May 22. PMID 31115918
- [Background] Norris CM, Close JCT. Prehabilitation for the Frailty Syndrome: Improving Outcomes for Our Most Vulnerable Patients. Anesth Analg. 2020 Jun;130(6):1524-1533. doi: 10.1213/ANE.0000000000004785. PMID 32384342
- [Background] Deiner S, Westlake B, Dutton RP. Patterns of surgical care and complications in elderly adults. J Am Geriatr Soc. 2014 May;62(5):829-35. doi: 10.1111/jgs.12794. Epub 2014 Apr 14. PMID 24731176
- [Background] Clegg A, Young J, Iliffe S, Rikkert MO, Rockwood K. Frailty in elderly people. Lancet. 2013 Mar 2;381(9868):752-62. doi: 10.1016/S0140-6736(12)62167-9. Epub 2013 Feb 8. PMID 23395245
- [Background] Panayi AC, Orkaby AR, Sakthivel D, Endo Y, Varon D, Roh D, Orgill DP, Neppl RL, Javedan H, Bhasin S, Sinha I. Impact of frailty on outcomes in surgical patients: A systematic review and meta-analysis. Am J Surg. 2019 Aug;218(2):393-400. doi: 10.1016/j.amjsurg.2018.11.020. Epub 2018 Nov 27. PMID 30509455
- [Background] Brown CH 4th, Max L, LaFlam A, Kirk L, Gross A, Arora R, Neufeld K, Hogue CW, Walston J, Pustavoitau A. The Association Between Preoperative Frailty and Postoperative Delirium After Cardiac Surgery. Anesth Analg. 2016 Aug;123(2):430-5. doi: 10.1213/ANE.0000000000001271. PMID 27096563
- [Background] Mahanna-Gabrielli E, Zhang K, Sieber FE, Lin HM, Liu X, Sewell M, Deiner SG, Boockvar KS. Frailty Is Associated With Postoperative Delirium But Not With Postoperative Cognitive Decline in Older Noncardiac Surgery Patients. Anesth Analg. 2020 Jun;130(6):1516-1523. doi: 10.1213/ANE.0000000000004773. PMID 32384341
- [Background] Watt J, Tricco AC, Talbot-Hamon C, Pham B, Rios P, Grudniewicz A, Wong C, Sinclair D, Straus SE. Identifying Older Adults at Risk of Delirium Following Elective Surgery: A Systematic Review and Meta-Analysis. J Gen Intern Med. 2018 Apr;33(4):500-509. doi: 10.1007/s11606-017-4204-x. Epub 2018 Jan 26. PMID 29374358
- [Background] McIsaac DI, Harris EP, Hladkowicz E, Moloo H, Lalu MM, Bryson GL, Huang A, Joanisse J, Hamilton GM, Forster AJ, van Walraven C. Prospective Comparison of Preoperative Predictive Performance Between 3 Leading Frailty Instruments. Anesth Analg. 2020 Jul;131(1):263-272. doi: 10.1213/ANE.0000000000004475. PMID 31569165
- [Background] Gleason LJ, Benton EA, Alvarez-Nebreda ML, Weaver MJ, Harris MB, Javedan H. FRAIL Questionnaire Screening Tool and Short-Term Outcomes in Geriatric Fracture Patients. J Am Med Dir Assoc. 2017 Dec 1;18(12):1082-1086. doi: 10.1016/j.jamda.2017.07.005. Epub 2017 Aug 31. PMID 28866353
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Morley JE, Malmstrom TK, Miller DK. A simple frailty questionnaire (FRAIL) predicts outcomes in middle aged African Americans. J Nutr Health Aging. 2012 Jul;16(7):601-8. doi: 10.1007/s12603-012-0084-2. PMID 22836700
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Darvall JN, Loth J, Bose T, Braat S, De Silva A, Story DA, Lim WK. Accuracy of the Clinical Frailty Scale for perioperative frailty screening: a prospective observational study. Can J Anaesth. 2020 Jun;67(6):694-705. doi: 10.1007/s12630-020-01610-x. Epub 2020 Mar 3. PMID 32128722
- [Background] Purdon PL, Sampson A, Pavone KJ, Brown EN. Clinical Electroencephalography for Anesthesiologists: Part I: Background and Basic Signatures. Anesthesiology. 2015 Oct;123(4):937-60. doi: 10.1097/ALN.0000000000000841. PMID 26275092
- [Background] Purdon PL, Pavone KJ, Akeju O, Smith AC, Sampson AL, Lee J, Zhou DW, Solt K, Brown EN. The Ageing Brain: Age-dependent changes in the electroencephalogram during propofol and sevoflurane general anaesthesia. Br J Anaesth. 2015 Jul;115 Suppl 1(Suppl 1):i46-i57. doi: 10.1093/bja/aev213. PMID 26174300
- [Background] Giattino CM, Gardner JE, Sbahi FM, Roberts KC, Cooter M, Moretti E, Browndyke JN, Mathew JP, Woldorff MG, Berger M; MADCO-PC Investigators. Intraoperative Frontal Alpha-Band Power Correlates with Preoperative Neurocognitive Function in Older Adults. Front Syst Neurosci. 2017 May 8;11:24. doi: 10.3389/fnsys.2017.00024. eCollection 2017. PMID 28533746
- [Background] Pedemonte JC, Plummer GS, Chamadia S, Locascio JJ, Hahm E, Ethridge B, Gitlin J, Ibala R, Mekonnen J, Colon KM, Westover MB, D'Alessandro DA, Tolis G, Houle T, Shelton KT, Qu J, Akeju O. Electroencephalogram Burst-suppression during Cardiopulmonary Bypass in Elderly Patients Mediates Postoperative Delirium. Anesthesiology. 2020 Aug;133(2):280-292. doi: 10.1097/ALN.0000000000003328. PMID 32349072
- [Background] Kaiser HA, Hirschi T, Sleigh C, Reineke D, Hartwich V, Stucki M, Rummel C, Sleigh J, Hight D. Comorbidity-dependent changes in alpha and broadband electroencephalogram power during general anaesthesia for cardiac surgery. Br J Anaesth. 2020 Oct;125(4):456-465. doi: 10.1016/j.bja.2020.06.054. Epub 2020 Jul 31. PMID 32747077
- [Background] Evered LA, Vitug S, Scott DA, Silbert B. Preoperative Frailty Predicts Postoperative Neurocognitive Disorders After Total Hip Joint Replacement Surgery. Anesth Analg. 2020 Nov;131(5):1582-1588. doi: 10.1213/ANE.0000000000004893. PMID 33079882
- [Derived] Boncompte G, Sun H, Elgueta MF, Benavides J, Carrasco M, Morales MI, Calderon N, Contreras V, Westover MB, Cortinez LI, Akeju O, Pedemonte JC. Intraoperative electroencephalographic marker of preoperative frailty: A prospective cohort study. J Clin Anesth. 2023 Jun;86:111069. doi: 10.1016/j.jclinane.2023.111069. Epub 2023 Feb 2. PMID 36738630

DOCUMENTS (2):
  • Statistical Analysis Plan (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT04783662/SAP_000.pdf
  • Informed Consent Form (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT04783662/ICF_001.pdf